CLINICAL TRIAL: NCT03154541
Title: SynRinse Irrigation Pilot (SIP) Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Greg Davis, Associate Professor, Otolaryngology - Head and Neck Surgery, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001280
Record Dates: First submitted 2017-05-03; First posted 2017-05-16 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Sinusitis, Chronic; Cystic Fibrosis With Other Manifestations
Keywords: Chronic Rhinosinusitis (CRS), Cystic Fibrosis related CRS
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-blinded single arm cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non Cystic Fibrosis (CF) cohort (Experimental): The first 10 non-CF subjects will be instructed to once daily irrigate both nasal passages with SynRinse (supplied) delivered via nasal irrigation using the NeilMed® Sinus Rinse™ system for 1 week. No prescription is necessary. The subjects will be asked to refrain from performing any sinus irrigations during the test treatment period with any product including saline.
  The second set of 10 non-CF subjects (if the study continues to this point) will be instructed to irrigate both nasal passages twice daily (rather than once daily) for one week with SynRinse (supplied). The subjects will be asked to refrain from performing any sinus irrigations during the test treatment period with any product including saline.
  Interventions: Drug: Synrinse
- Cystic Fibrosis (CF) cohort (Experimental): The first 5 subjects in the CF cohort will irrigate with with SynRinse delivered via nasal irrigation using the NeilMed Sinus Rinse system for 1 week. The second set of 5 subjects with CF will irrigate both nasal passages twice daily for one week with SynRinse.
  Interventions: Drug: Synrinse

INTERVENTIONS:
Drug: Synrinse — Non-CF Cohort The first 10 non-CF subjects will be instructed to once daily irrigate both nasal passages with SynRinse (supplied) delivered via nasal irrigation using the NeilMed® Sinus Rinse™ system for 1 week. The subjects will be asked to refrain from performing any sinus irrigations during the test treatment period with any product including saline.
  The second set of 10 non-CF subjects (if the study continues to this point) will be instructed to irrigate both nasal passages twice daily (rather than once daily) for one week with SynRinse (supplied). The subjects will be asked to refrain from performing any sinus irrigations during the test treatment period with any product including saline.
  CF Cohort The first 5 subjects in the CF cohort will irrigate with with SynRinse delivered via nasal irrigation using the NeilMed Sinus Rinse system for 1 week. The second set of 5 subjects with CF will irrigate both nasal passages twice daily for one week with SynRinse.

SUMMARY:
Assess if the use of SYNRINSE can improve short-term subjective and objective outcome measures after one week in patients with active Chronic Rhinosinusitis (CRS) who have had prior sinus surgery.

DETAILED DESCRIPTION:
SYNRINSE is osmotically balanced and also contains soluble chitosan-argininamide, a modified natural glycopolymer that has a number of properties important to relieving the symptoms of mucus build up and bacterial biofilms. First, SYNRINSE reduces the viscosity of biofilms, the protective environment of infective bacteria that prevents topical antibiotics and other rinses to penetrate to reach the bacterial. By disrupting biofilms, SYNRINSE allows them to be cleared from the sinuses. Second, SYNRINSE has been shown to interact with the polymers comprise mucus, loosening thick, sticky layers and reducing their ability to adhere together and to mucosal surfaces. Third, all of the components in SYNRINSE are biocompatible and soothing to sensitive nasal cavities.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* Meet diagnostic criteria for CRS (as defined by the AAO-HNS 2015 Clinical Practice Guidelines for Adult Sinusitis).
* Have undergone at least one functional endoscopic sinus surgery, be at least 6 weeks out from surgery, be free of any complication from surgery, and have patent sinuses confirmed by nasal endoscopy.
* Have active sinus disease as defined as purulent sinus discharge visualized on nasal endoscopy.
* Have more than mild symptoms as determined by the SNOT-22 with a score >20.
* Be willing to hold off on standard therapy for chronic sinusitis for 1 week including oral antibiotics and/or oral steroids.
* If on topical steroids for greater than 1 month (sprays, drops, or irrigation) these will be continued based on the patients' current use (continued if they are already on them, not initiated if they are not on them).
* Must be able to irrigate with large volume/low pressure nasal lavage throughout the study.

Exclusion Criteria

:• Have an allergy to shell fish.

* Be able to return for follow up evaluation in 1 week (+ up to 5 days if needed)
* Have obstructive nasal polyps
* Participants who have used topical antibiotics within 4 weeks of treatment or are actively using them and unwilling to stop
* Participants who have used systemic steroids within 4 weeks of treatment
* Are unable to give informed consent or complete self-administered questionnaires written in English because of cognitive impairment, language barrier, or severe medical conditions.
* Have a terminal illness or significant immune dysfunction.
* Have severe or emergent complications from CRS or presence of a sinus tumor.
* Patients with Cystic Fibrosis will be recruited in a parallel study.
* Participants who are unwilling to discontinue other sinus irrigations treatments and steroid lavage if already on them (including baby shampoo, surfactant, colloid silver, manuka honey, iodine, alcohol, tea tree oil, or any other compound).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Sino-Nasal Outcome Test 22 (SNOT-22) | 1 week
  Test pre-treatment SNOT-22 (sinusitis-specific quality of life) and compare to post-treatment SNOT-22 scores to measure any change in disease specific quality of life.

SECONDARY OUTCOMES:
Sinus bacteria culture | 1 week
  Obtain a pre-treatment endoscopic collected culture and a post-treatment endoscopic collected culture to see if the treatment impacts a pathogen detected in the pre-treatment culture.
Lund-Kennedy Endoscopy Score (LKES) | 1 week
  Measure change in pre-treatment LKES and post-treatment LKES to determine if treatment impacts any change in the appearance of the patient's sinuses on endoscopy
Visual Analog Scale (VAS) | 1 week
  Determine the tolerability of SYNRINSE as measured on a 10cm VAS
Future use questionnaire | 1 week
  Record percentage of subjects willing to use SYNRINSE in the future

CONTACTS AND LOCATIONS:
Overall Officials: Greg Davis, MD, Principal Investigator — UW
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No